CLINICAL TRIAL: NCT00456391
Title: The Utility of Performing Brain CT Scan in Non Trauma Patients at the Pediatric Emergency Unit. A Retrospective Observational Study.
Brief Title: The Utility of Performing Brain CT Scan in Non Trauma Patients at the Pediatric Emergency Unit
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Other Study IDs: 5200906.EMC
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Convulsions; Increased Intracraneal Pressure
Keywords: Brain CT scan; Pediatric emergency room
MeSH Terms: conditions — Seizures | interventions — Health Records, Personal

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Medical history
Procedure: Brain CT scan

SUMMARY:
Pediatric patients are admitted to the emergency room for diverse causes, beside trauma, patients can present with convulsions, suspicion of brain tumor or increased intracranial pressure. In most of the cases a brain CT is performed even before physical examination by a skilled neurologist. The amount of radiation that the children are exposed is equivalent to 100 plain chest X rays. The purpose of this tudy is to examinate in a retrospective study what were the indications for CT study and what was the incidence of relevant abnormal findings that required emergency intervention or referral.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the pediatric age that underwent brain CT scan in the pediatric emergency room

Exclusion Criteria:

* Patients with recent history of trauma

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2006-10; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Study Director — Pediatric Hematology Unit, Ha'Emek Medical Center; Waheeb Sakran, MD, Principal Investigator — Pediatric Dpt B - Ha'Emek Medical Center; Izat Hatib, MD, Principal Investigator — Pediatric Dpt B - Ha'Emek Medical Center
Locations (1):
- Pediatric Dpt B and Pediatric Emergency Room - HaEmek Medical Center, Afula, Israel